CLINICAL TRIAL: NCT03764891
Title: Far Eastern Memorial Hospital
Brief Title: Clinical Outcomes of Transvaginal Mesh Procedures for Cystocele Repair: Comparisons of Uphold and Perigee Systems
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 107159-E
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Organ Prolapse; Surgical Mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uphold: Patients who underwent Uphold procedure
  Interventions: Procedure: Uphold
- Perigee: Patients who underwent Perigee procedure
  Interventions: Procedure: Perigee

INTERVENTIONS:
Procedure: Uphold — Uphold system in treating women with cystocele
  Groups: Uphold
Procedure: Perigee — Perigee system in treating women with cystocele
  Groups: Perigee

SUMMARY:
Pelvic organ prolapse (POP) is a major health concern, affecting more than 30% of women.

The aim of this study was to compare the clinical outcomes of Uphold system and Perigee system in treating women with cystocele.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is a major health concern, affecting more than 30% of women. Traditional vaginal surgery with native tissue is associated with high recurrence rate. Thus, synthetic meshes were introduced into POP surgery and became the mainstream. Several transvaginal mesh procedures, such as Uphold system (Boston Scientific) and Perigee system (American Medical Systems Inc), have been used for cystocele repair. Perigee system is a trans-obturator four-arm mesh device attached to proximal and distal arcus tendineus fasciae pelvis. Nonetheless, Uphold system, is a single incised, two-arm anterior sacrospinous mesh fixation system. Both systems can be used for cystocele repair, despite Uphold system can be used for concomitant repair of apical prolapse. The aim of this study was to compare the clinical outcomes of Uphold system and Perigee system in treating women with cystocele.

ELIGIBILITY:
Inclusion Criteria:

1. Vaginal anterior wall prolapse greater than or equal to second phase of POP-Q
2. Underwent Uphold or Perigee procedures

Exclusion Criteria:

* nil

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pelvic organ prolapse patients underwent Uphold or Perigee surgeries
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of pelvic organ prolapse | 10 year
  Compare the recurrence rate of Uphold system and Perigee system in treating women with cystocele.

SECONDARY OUTCOMES:
Complication rate | 10 years
  Compare the complication rate (such as mesh extrusion, dyspareunia, pelvic pain, voiding difficult, etc) of Uphold system and Perigee system in treating women with cystocele.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan